CLINICAL TRIAL: NCT03386838
Title: A Randomized, Global, Open-label Study of Nivolumab in Combination With BMS-986205 vs Standard of Care EXTREME Regimen in First-line Recurrent/Metastatic Squamous Cell Carcinoma of Head and Neck
Brief Title: An Immuno-therapy Study of Nivolumab in Combination With Experimental Medication BMS-986205 Compared to Standard of Care EXTREME Regimen in First-line Recurrent/Metastatic Squamous Cell Carcinoma of Head and Neck
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA017-063; 2017-003059-46 (EudraCT Number)
Record Dates: First submitted 2017-12-22; First posted 2017-12-29 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab; linrodostat; Cetuximab; Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab and BMS-986205 (Experimental): Nivolumab administered in combination with BMS-986205
  Interventions: Biological: Nivolumab; Drug: BMS-986205
- EXTREME study regimen (Active Comparator): Cetuximab + Cisplatin/Carboplatin + Fluorouracil
  Interventions: Biological: Cetuximab; Drug: Cisplatin; Drug: Carboplatin; Drug: Fluorouracil

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Nivolumab and BMS-986205
Drug: BMS-986205 — Administered 100mg orally once daily for a maximum of 104 weeks
  Arms: Nivolumab and BMS-986205
Biological: Cetuximab — 400 mg/m² intravenous administration once only, then 250 mg/m² weekly maintenance until disease progression, unacceptable toxicity, withdrawal of informed consent, or other reason
  Arms: EXTREME study regimen
Drug: Cisplatin — Cisplatin (100 mg/m2) every 3 weeks (Up to 6 cycles)
  Arms: EXTREME study regimen
Drug: Carboplatin — Carboplatin (AUC of 5 mg per milliliter per minute) every 3 weeks (Up to 6 cycles)
  Arms: EXTREME study regimen
Drug: Fluorouracil — 1000 mg/m² per day for 4 days, every 3 weeks (Up to 6 cycles)
  Arms: EXTREME study regimen

SUMMARY:
This is a study of Nivolumab in combination with experimental medication BMS-986205 compared to the standard of care EXTREME regimen in head and neck cancer that has come back after initial treatment, or is widespread when first diagnosed.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck (SCCHN), from any of the following primary sites only: oral cavity, oropharynx, hypopharynx, and larynx.
* Recurrent or metastatic disease that is not amenable to therapy with curative intent (surgery or radiation therapy with or without chemotherapy)
* No prior treatment with systemic anti-cancer therapy for SCCHN, unless protocol specified criteria are met
* ECOG Performance Status of 0-1
* Measurable disease by CT or MRI per RECIST 1.1 criteria

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Recurrent or metastatic carcinoma of the nasopharynx, squamous cell carcinoma of unknown primary, squamous cell carcinoma that originated from the skin and salivary gland or paranasal sinus, non-squamous histologies (eg, mucosal melanoma)
* Participants with untreated CNS metastases are excluded
* Participants with carcinomatous meningitis
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as determined by Blinded Independent Central Review (BICR) using RECIST 1.1 | Approximately 2 years
Overall survival (OS) | Approximately 40 months
Objective response rate (ORR) determined by BICR using RECIST 1.1 | Approximately 2 years

SECONDARY OUTCOMES:
Number of adverse events (AE) | Approximately 2 years
Number of serious adverse events (SAE) | Approximately 2 years
Time to meaningful symptomatic deterioration (TTSD) | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx